CLINICAL TRIAL: NCT05026411
Title: Assessment of Food Reward Circuit Change in Individuals Receiving Orthodontic Treatment With Diffusion Tensor Imaging
Brief Title: Food Reward Circuit Change by Orthodontics
Acronym: DTI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Muğla Sıtkı Koçman University (Other); The Scientific and Technological Research Council of Turkey (Other); Balikli greek hospital foundation (Unknown)
Responsible Party: Principal Investigator, Banu Kılıç, Assistant Professor, Bezmialem Vakif University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: bkilic002; 119S125 (Other Grant/Funding Number: THE SCIENTIFIC AND TECHNOLOGICAL RESEARCH COUNCIL OF TURKEY)
Record Dates: First submitted 2021-04-01; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Eating Disorders; Eating Behavior; Eating Habit; Orthodontic Appliance Complication
MeSH Terms: conditions — Feeding and Eating Disorders; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Diffusion tensor imagings will be taken from the patients at the beginning of the orthodontic treatment, in the first year of treatment and 6 months after the treatment ends.
Masking Description: The radiologist will be blinded to who the films are from and at what stage of the treatment they were taken.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orthodontic patients (Other): Magnetic resonance images will be taken from 20 individuals with eating disorders before fixed orthodontic treatment, 12 months of orthodontic treatment and 6 months after orthodontic treatment finished
  Interventions: Diagnostic Test: T 0 Diffusion Tensor MR; Diagnostic Test: T 1 Diffusion Tensor MR; Diagnostic Test: T 2 Diffusion Tensor MR

INTERVENTIONS:
Diagnostic Test: T 0 Diffusion Tensor MR — Magnetic resonance images has been taken from 20 individuals with eating disorders before fixed orthodontic treatment
Diagnostic Test: T 1 Diffusion Tensor MR — Magnetic resonance images will be taken from 20 individuals with eating disorders after 12 months of orthodontic treatment.
Diagnostic Test: T 2 Diffusion Tensor MR — Magnetic resonance images will be taken from 20 individuals with eating disorders 6 months after orthodontic treatment finished

SUMMARY:
It has been described in obese individuals in which decreased basal metabolism as well as dopaminergic changes in the prefrontal cortex and striatum parallels the increased activation of reward brain regions in response to delicious food cues. Our aim is to explore different neurobehavioral dimensions of food choices and motivational processes in the light of this information, and to reveal whether these behaviors can be changed by operant conditioning with neuroimaging methods for phenotypes at risk.

DETAILED DESCRIPTION:
The incidence of eating disorders in society is increasing day by day and is becoming an increasingly serious problem. Overweight people are suggested to exhibit eating behavior to cope with anxiety, depressed mood, anger and other negative emotions. Studies in humans and animals have shown that obesity is associated with changes in dopaminergic neurotransmission. Changes in brain locations associated with satiety and hunger centers (hypothalamus, hippocampal gyrus, amygdala, insula, cerebellum and midbrain) of obese patients have been shown. It has been reported that cognitive control strategies that can lead to more effective impulse control behaviors should be applied for obesity treatment, which is considered as an addiction in which food is perceived as a reward nowadays.

During the first week of fixed orthodontic treatment, all the patients have pain and various discomforts with food, and after each appointment, the pain occurs while chewing. Patients declare having prolonged eating times due to difficulty in chewing, food impaction under the brackets and complains about not being able to consume sugar-containing foods due to maintain oral hygen. It is known that individuals who have eating disorders have a disturbance in their food rewarding properties and eating behavior. They eat in response to emotions rather than to meet energy needs. Pharmacological and bariatric surgical interventions are more successful than dietary lifestyle interventions because these interventions reduced not only the hunger but also the reward value of the homeostatic and hedonic brain regions of the foods. However, there is no study of whether enjoying from the food, perceiving food as a reward or individuals eating habits can be changed. The hypothesis of this study is that as a result of orthodontic treatment in which individuals experience negative emotions during each meal for two years there will be a change in the way of individuals' interpretation of food.

In order to investigate this hypothesis, eating attitudes and eating habit questionnaires will be applied to healthy volunteers with a body mass index of 25 and above chosen from patients who applied to our clinic for fixed orthodontic treatment. Thus, individuals with emotional eating, externally induced eating, restrained eating disorders and eating habits of these individuals will be identified. Magnetic resonance images will be taken from 20 individuals with eating disorders before fixed orthodontic treatment, 12 months of orthodontic treatment and 6 months after orthodontic treatment finished. By means of magnetic resonance imaging (MRI) and diffusion tensor imaging (DTG), the microstructural changes in axonal and myelin structures in the tracts of the selected appetite and satiety centers in the brain will be defined. The presence of changes by the orthodontic treatment in nutritional perceptions will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Patients thought to have emotional eating, restrained eating and external eating.
2. patients between the ages of 18-60
3. Patients with minor to moderate crowding in the mandibular and maxillary arches not exceeding 7 mm
4. Orthodontic patients who need to be treated with fixed treatment without extraction.
5. Class 1 healthy patients according to the American Society of Anesthesiologists (ASA) criteria 20 individuals selected from amongst will constitute our main sample group.

Exclusion Criteria:

1. Maxillary expansion apparatus, transpalatal arch, Herbst, Forsus etc. before fixed treatment. Patients who require fixed non-treatment devices such as fixed devices will not be included in the study.
2. Patients who require constant use of devices containing materials that may contain steel other than tubes and brackets as orthodontic materials will not be included.
3. Although it could not be detected at the beginning of the treatment if any of the treatment methods (extraction, etc.) other than the standardized protocol are required in the future, the patient will be excluded from the study.
4. Before the patients start orthodontic treatment, a consultation will be requested from the Department of Mental Health and Diseases and the patients who are not found suitable will be excluded from the study by the initiative of the psychiatrist who examines the patient without asking a reason for the doctor-patient confidentiality.
5. Before the patients start orthodontic treatment, a consultation will be requested from the dietician and the patients who are not found suitable will be excluded from the study by the initiative of the dietician who examines the patient without asking a reason for the doctor-patient confidentiality.
6. Before the patients start orthodontic treatment, a consultation will be requested from the internal medicine doctor if there is any doubt that there may be an organic basis for patients to have a high BMI. The patients who are not found suitable will be excluded from the study by the initiative of the internal medicine doctor who examines the patient without asking a reason for the doctor-patient confidentiality.
7. Patients using medical treatment due to a known disease before orthodontic treatment will be excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
T0 -T1 DTMR fractional anisotropy change | 12 months
  The microstructural changes in axonal and myelin structures in the tracts of the selected appetite and satiety centers in the brain will be defined. Fractional anisotropy, apparent diffusion coefficient, mean diffusivity and radial diffusivity parameters from different localizations will be measured. A hierarchical cluster analysis will be performed for centers with differing tensor imaging measurement values and a heatmap will be drawn according to the measurement level, and the brain centers with the most statistically significant difference will be scored and listed. All analyzes will be presented by using open source R packages by visualizing them with the help of tables and graphs. The written codes will be made available to everyone on open source sharing pages (such as github, bitbucket)
T1-T2 DTMR fractional anisotropy change | 6 months after the end of fixed orthodontic treatment
  The microstructural changes in axonal and myelin structures in the tracts of the selected appetite and satiety centers in the brain will be defined after orthodontic treatment. Fractional anisotropy parameters from different localizations will be measured. A hierarchical cluster analysis will be performed for centers with differing tensor imaging measurement values and a heatmap will be drawn according to the measurement level, and the brain centers with the most statistically significant difference will be scored and listed. All analyzes will be presented by using open source R packages by visualizing them with the help of tables and graphs. The written codes will be made available to everyone on open source sharing pages (such as github, bitbucket)
T0 -T1 DTMR apparent diffusion coefficient change | 12 months
  The microstructural changes in axonal and myelin structures in the tracts of the selected appetite and satiety centers in the brain will be defined. Apparent diffusion coefficient parameters from different localizations will be measured. A hierarchical cluster analysis will be performed for centers with differing tensor imaging measurement values and a heatmap will be drawn according to the measurement level, and the brain centers with the most statistically significant difference will be scored and listed. All analyzes will be presented by using open source R packages by visualizing them with the help of tables and graphs. The written codes will be made available to everyone on open source sharing pages (such as github, bitbucket)
T1-T2 DTMR Apparent diffusion coefficient change | 6 months
  The microstructural changes in axonal and myelin structures in the tracts of the selected appetite and satiety centers in the brain will be defined after orthodontic treatment. Apparent diffusion coefficient parameters from different localizations will be measured. A hierarchical cluster analysis will be performed for centers with differing tensor imaging measurement values and a heatmap will be drawn according to the measurement level, and the brain centers with the most statistically significant difference will be scored and listed. All analyzes will be presented by using open source R packages by visualizing them with the help of tables and graphs. The written codes will be made available to everyone on open source sharing pages (such as github, bitbucket)
T0 -T1 DTMR mean diffusivity change | 12 months
  The microstructural changes in axonal and myelin structures in the tracts of the selected appetite and satiety centers in the brain will be defined. Mean diffusivity parameters from different localizations will be measured. A hierarchical cluster analysis will be performed for centers with differing tensor imaging measurement values and a heatmap will be drawn according to the measurement level, and the brain centers with the most statistically significant difference will be scored and listed. All analyzes will be presented by using open source R packages by visualizing them with the help of tables and graphs. The written codes will be made available to everyone on open source sharing pages (such as github, bitbucket)
T1-T2 DTMR mean diffusivity change | 6 months
  The microstructural changes in axonal and myelin structures in the tracts of the selected appetite and satiety centers in the brain will be defined after orthodontic treatment. Mean diffusivity change parameters from different localizations will be measured. A hierarchical cluster analysis will be performed for centers with differing tensor imaging measurement values and a heatmap will be drawn according to the measurement level, and the brain centers with the most statistically significant difference will be scored and listed. All analyzes will be presented by using open source R packages by visualizing them with the help of tables and graphs. The written codes will be made available to everyone on open source sharing pages (such as github, bitbucket)
T0 -T1 DTMR Radial diffusivity change | 12 months
  The microstructural changes in axonal and myelin structures in the tracts of the selected appetite and satiety centers in the brain will be defined. Radial diffusivity parameters from different localizations will be measured. A hierarchical cluster analysis will be performed for centers with differing tensor imaging measurement values and a heatmap will be drawn according to the measurement level, and the brain centers with the most statistically significant difference will be scored and listed. All analyzes will be presented by using open source R packages by visualizing them with the help of tables and graphs. The written codes will be made available to everyone on open source sharing pages (such as github, bitbucket)
T1-T2 DTMR radial diffusivity change | 6 months
  The microstructural changes in axonal and myelin structures in the tracts of the selected appetite and satiety centers in the brain will be defined after orthodontic treatment. Radial diffusivity parameters from different localizations will be measured. A hierarchical cluster analysis will be performed for centers with differing tensor imaging measurement values and a heatmap will be drawn according to the measurement level, and the brain centers with the most statistically significant difference will be scored and listed. All analyzes will be presented by using open source R packages by visualizing them with the help of tables and graphs. The written codes will be made available to everyone on open source sharing pages (such as github, bitbucket)

SECONDARY OUTCOMES:
T0-T1 Dutch Eating Behaviour Questionnaire Score Change | 12 months
  33 items, which measures emotional (13 items), external, and restrained eating (both 10 items) rated on a five-point scale from 1 (never) to 5 (very often) will be evaluated.
  The presence of changes at eating behaviour by the orthodontic treatment in nutritional perceptions will be measured. A decrease in DEBQ scores will be perceived as a positive improvement.
T1-T2 Dutch Eating Behaviour Questionnaire Score Change | 6 months after the end of fixed orthodontic treatment
  33 items, which measures emotional (13 items), external, and restrained eating (both 10 items) rated on a five-point scale from 1 (never) to 5 (very often) will be evaluated.
  If there is a presence of changes at eating behavior by the orthodontic treatment we will be able to measure if they are stable or not. A decrease in DEBQ scores or a stabilization of the dropped score will be perceived as a positive development.
T0-T1 Eating Attitude Test Score Change | 12 months
  It includes 40 items in which the frequencies of attitudes and beliefs are rated using 6-point scale. A score of 30 and above is commonly used as a cut-off point to identify individuals with anorexia or bulimia. The presence of changes at eating attitude by the orthodontic treatment in nutritional perceptions will be measured. A decrease in Eating Attitude Test scores will be perceived as a positive development.
T1-T2 Eating Attitude Test Score Change | 6 Months
  It includes 40 items in which the frequencies of attitudes and beliefs are rated using 6-point scale. A score of 30 and above is commonly used as a cut-off point to identify individuals with anorexia or bulimia. If there is a presence of changes at eating attitude by the orthodontic treatment we will be able to measure if they are stable or not. Eating Attitude Test scors falling or remaining stable will be perceived as a positive development.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Kılıç, Study Director — Bezmialem Vakif University
Locations (1):
- Banu Kilic, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bozan N, Bas M, Asci FH. Psychometric properties of Turkish version of Dutch Eating Behaviour Questionnaire (DEBQ). A preliminary results. Appetite. 2011 Jun;56(3):564-6. doi: 10.1016/j.appet.2011.01.025. Epub 2011 Jan 26. PMID 21277923
- [Background] Kroemer NB, Small DM. Fuel not fun: Reinterpreting attenuated brain responses to reward in obesity. Physiol Behav. 2016 Aug 1;162:37-45. doi: 10.1016/j.physbeh.2016.04.020. Epub 2016 Apr 13. PMID 27085908
- [Background] Alkan A, Sahin I, Keskin L, Cikim AS, Karakas HM, Sigirci A, Erdem G. Diffusion-weighted imaging features of brain in obesity. Magn Reson Imaging. 2008 May;26(4):446-50. doi: 10.1016/j.mri.2007.10.004. Epub 2007 Dec 11. PMID 18063337
- [Background] Garcia-Garcia I, Horstmann A, Jurado MA, Garolera M, Chaudhry SJ, Margulies DS, Villringer A, Neumann J. Reward processing in obesity, substance addiction and non-substance addiction. Obes Rev. 2014 Nov;15(11):853-69. doi: 10.1111/obr.12221. Epub 2014 Sep 29. PMID 25263466
- [Background] Sergl HG, Klages U, Zentner A. Pain and discomfort during orthodontic treatment: causative factors and effects on compliance. Am J Orthod Dentofacial Orthop. 1998 Dec;114(6):684-91. doi: 10.1016/s0889-5406(98)70201-x. PMID 9844209